CLINICAL TRIAL: NCT06789198
Title: FusionVAC22_02: DNAJB1-PRKACA Fusion Transcript-based Peptide Vaccine for Fibrolamellar Hepatocellular Carcinoma Patients and Other Tumor Entities Carrying the Oncogenic Driver Fusion
Brief Title: Peptide Vaccine for Fibrolamellar Hepatocellular Carcinoma Patients and Other Tumor Entities Carrying the Driver Fusion DNAJB1-PRKACA
Acronym: FusionVAC22_02
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FusionVAC22_02; 2024-519387-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Fibrolamellar Hepatocellular Carcinoma (FLC)
Keywords: DNAJB1-PRKACA fusion transcript; Fibrolamellar hepatocellular carcinoma (FL-HCC)
MeSH Terms: conditions — Fibrolamellar hepatocellular carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial conduction (Experimental): All trial participants will recieve at least two vaccinations with Fusion-VAC-XS15 and one optional boster vaccination depending on the T-cell response
  Interventions: Drug: Vaccination of Fusion-VAC-XS15

INTERVENTIONS:
Drug: Vaccination of Fusion-VAC-XS15 — FusionVAC-22 peptide will be administered subcutaneously (s.c.) with the TLR1/2 ligand XS15 (50 µg) emulsified in Montanide ISA 51 VG (1:1).
  A total of two vaccinations are planned, 4 weeks apart from each other. If no sufficient T cell response is achieved at the end of treatment visit (28 days after last vaccination) a booster vaccination at day 56 (+7 days) after the second vaccination can be applied

SUMMARY:
The aim of this clinical trial is to evaluate the immunogenicity along with safety and toxicity as well as first efficacy of a DNAJB1-PRKACA fusion transcript-based peptide vaccine (Fusion-VAC-XS15) in patients with FL-HCC or other cancer entities carrying the DNAJB1-PRKACA fusion transcript as adjuvant treatment

DETAILED DESCRIPTION:
To date, beyond surgery, there are no approved drugs and no standard of care for the treatment of FLC patients. Relapse rates after remission inducing therapies (surgery, radiation, liver transplant, systemic therapy approaches) are very high. With FusionVAC-XS15 the sponsor aims to activate the immune system specifically against the gene fusion to eradicate remaining tumor cells to improve disease remission and finally enable long-term disease-free survival.

Patients with confirmed diagnosis of FL-HCC or other cancer entities carrying the DNAJB1-PRKACA fusion transcript and fulfilling the below outlined inclusion criteria will be enrolled into the clinical trial. The trial population will consist of both genders. Gender distribution in the trial is supposed to reflect the distribution in the real patient population; there will be no a priori defined quantitative ratio between females and males. FusionVAC-22 peptide will be administered subcutaneously (s.c.) with the TLR1/2 ligand XS15 (50 µg) emulsified in Montanide ISA 51.

A total of two vaccinations are planned, 4 weeks apart from each other. If no sufficient T cell response is achieved at the end of treatment visit (28 days after last vaccination) a booster vaccination at day 56 (+7 days) after the second vaccination can be applied

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent document.
* Histologically confirmed Fibrolamellar hepatocellular carcinoma (FL-HCC) or other malignant disease in an adjuvant setting, defined as:

  * Presence of DNAJB1-PRKACA fusion transcript, assessed by RNA-based NGS or RT-PCR
  * Achievement of complete remission (CR) according to RECIST1.1 by any of the following therapeutic measures:
* surgical procedures,
* radiotherapy,
* local therapeutic measures (e.g. TACE, SIRT, etc.)
* systemic treatment (e.g. chemotherapy)
* Age ≥ 12 years. Note: Subjects aged ≥ 12 years but < 18 are eligible to enroll only after 6 adult patients have been enrolled in the study.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Adequate laboratory values for

  * Absolute Lymphocyte Count > 500 /µl
  * Platelets > 50.000 /µl
  * Creatinine clearance GFR > 30 ml/min
  * Alanine aminotransferase (ALT) and aminotransferase (AST) ≤ 5 times upper limit range
  * Bilirubin ≤ 3 mg/dl
* Negative serological hepatitis B test or negative PCR in case of positive serological test without evidence of an active infection, negative testing of hepatitis C RNA, negative HIV test within 6 weeks prior to study inclusion.
* Female patients of child bearing potential (FCBP) and male patients with partners of child bearing potential who are sexually active must agree to the use of two effective forms (at least one highly effective method) of contraception. This should be started from the signing of the informed consent and be continued until 3 months (both female and male patients) after last dose of the vaccination
* For FCBP two negative pregnancy tests (sensitivity of at least 25 mIU/mL) prior to first application of the study drug (vaccination at visit V1), one at screening and the other one at visit V1 prior (< 24h) to first vaccination.
* Postmenopausal or evidence of non-child-bearing status.
* Be willing to minimize blood and body fluid exposure after vaccination until end of study

  * Refrain from sperm or ovary egg donation
  * Refrain from blood donation

Exclusion Criteria:

* Pregnant or breastfeeding.
* Unwilling or unable to follow the study schedule for any reason.
* Concurrent or previous treatment within 14 days in another interventional clinical trial with an investigational anti-cancer treatment.
* Concurrent treatment with any of the following therapeutic measures:

  * surgical procedures,
  * radiotherapy,
  * local therapeutic measures (e.g. TACE, SIRT, etc.)
  * systemic treatment (e.g. chemotherapy)
* Concurrent or previous treatment within 6 months with an anti-cancer vaccine treatment.
* Any live vaccine therapy used for prevention of infectious diseases within 28 days of study treatment
* Known sensitivity to or history of allergic reactions to investigational drug.
* Active autoimmune disease that has required systemic treatment in the past 2 years, or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids (> 10 mg per day) or immunosuppressive agents (Please note, patients after liver transplantation requiring immunosupressants are allowed).
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy of vaccination | until 84 days after second vaccination
  Primary objectives of the planned trial are to assess immunogenicity in terms of induction of peptide specific T-cell responses
Safety of the vaccination | from first vaccination until 12 months after last vaccination
  Primary objective of the planned trial is to assess safety and toxicity of the peptide vaccine. The safety and toxicity of the DNAJB1-PRKACA fusion transcript-based peptide vaccine is determined based on the Common Terminology Criteria for Adverse Events (CTCAE V 5.0) and assessed in a descriptive manner.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Tuebingen, Tübingen
  - Universitätsklinikum Tübingen, Kinderheilkunde I, Tübingen

IPD SHARING:
Plan to Share IPD: No